CLINICAL TRIAL: NCT00856284
Title: A Multicenter, Randomized, Double-Blind, Active-Controlled Study to Evaluate the Durability of the Efficacy and Safety of Alogliptin Compared to Glipizide When Used in Combination With Metformin in Subjects With Type 2 Diabetes
Brief Title: Efficacy and Safety of Alogliptin Plus Metformin Compared to Glipizide Plus Metformin in Patients With Type 2 Diabetes Mellitus
Acronym: ENDURE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SYR-322_305; 2008-007444-34 (Registry Identifier: EudraCT); U1111-1111-7397 (Registry Identifier: WHO); HKCTR-862 (Registry Identifier: HKUCTR); DOH-27-0709-2825 (Registry Identifier: SANCTR); 09/H0703/66 (Registry Identifier: NRES); NMRR-09-203-3590 (Registry Identifier: NMRR)
Record Dates: First submitted 2009-03-04; First posted 2009-03-05 (Estimated); Results first posted 2013-12-03 (Estimated); Last update posted 2013-12-03 (Estimated); Status verified 2013-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes Mellitus; Drug Therapy; Hyperinsulinism; Hyperglycemia; Glucose Intolerance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Hyperinsulinism; Hyperglycemia; Glucose Intolerance | interventions — alogliptin; Metformin; Glipizide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Metformin + Alogliptin 12.5 mg (Experimental): Alogliptin 12.5 mg, tablets, orally, once daily and the maximum tolerated dose of metformin (1500 mg to 3300 mg daily) for up to 104 weeks.
  Interventions: Drug: Alogliptin; Drug: Metformin
- Metformin + Alogliptin 25 mg (Experimental): Alogliptin 25 mg, tablets, orally, once daily and the maximum tolerated dose of metformin (1500 mg to 3300 mg daily) for up to 104 weeks.
  Interventions: Drug: Alogliptin; Drug: Metformin
- Metformin + Glipizide (Active Comparator): Glipizide 5 mg, tablets, orally, once daily and the maximum tolerated dose of metformin (1500 mg to 3300 mg daily) for up to 104 weeks. After at least 2 weeks of treatment but prior to Week 20, participants with persistent hyperglycemia (fasting plasma glucose ≥250 mg/dL) underwent a dose titration of glipizide up to 20 mg in 5-mg increments in 4-week intervals.
  Interventions: Drug: Metformin; Drug: Glipizide

INTERVENTIONS:
Drug: Alogliptin — Alogliptin tablets
  Other Names: SYR-322; Nesina
  Arms: Metformin + Alogliptin 12.5 mg; Metformin + Alogliptin 25 mg
Drug: Metformin — Metformin tablets
  Other Names: Glucophage
Drug: Glipizide — Glipizide tablets
  Other Names: Glucotrol
  Arms: Metformin + Glipizide

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of adding alogliptin, once daily (QD), compared to glipizide with metformin in diabetic patients.

DETAILED DESCRIPTION:
For patients diagnosed with type 2 diabetes mellitus, metformin is the usual first-line therapy in addition to diet control and exercise. For those patients with inadequate glycemic control with metformin monotherapy or experiencing serious side effects of metformin, sulfonylurea is a popular choice as a second-line oral antidiabetic treatment.

Alogliptin is a dipeptidyl peptidase-4 inhibitor currently being developed by Takeda for use in patients with type 2 diabetes mellitus.

This study is designed to further explore the durability of efficacy and safety of alogliptin compared to glipizide in type 2 diabetes mellitus patients whose blood sugar level is inadequately controlled with metformin therapy.

The duration of this study will be approximately 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Has a diagnosis of type 2 diabetes mellitus.
* Must meet one of the following:

  * Has been inadequately controlled on a stable daily dose of ≥1500 mg (or documented maximum tolerated dose) of metformin for at least 2 months prior to Screening.
  * Has been inadequately controlled (as defined by a glycosylated hemoglobin 7.5 - 10%, inclusive) on metformin <1500 mg without documented maximum tolerated dose.
* No treatment with antidiabetic agents other than metformin within 2 months prior to Screening (for Schedule A)/Pre-Screening (for Schedule B).
* Has body mass index within 23 kg/m^2 and 45 kg/m^2 unless the patient is Asian or of Asian descent, for whom the allowable body mass index will be ≥ 20 kg/m^2 and ≤ 35 kg/m^2, inclusive.
* Has fasting C-peptide concentration at least 0.8 ng.
* If regularly using non-excluded medications, must be on a stable dose at least 4 weeks prior to Screening/Pre-screening.
* Females of childbearing potential who are sexually active must agree to use adequate contraception, and can neither be pregnant, lactating or intends to donate ova from Screening throughout the duration of the study.
* Must be able and willing to monitor their blood glucose concentrations with a home monitor, and comply with protocol requirements including scheduled clinic appointments.

Exclusion Criteria:

* Systolic blood pressure greater than or equal to 150 mmHg and/or diastolic pressure greater than or equal to 90.
* Hemoglobin less than or equal to 12 g/dL for males and less than or equal to 10 g/dL for females at Screening Visit.
* Alanine aminotransferase greater than or equal to 2.5 times the upper limit of normal at Screening Visit.
* Serum creatinine greater than or equal to 1.5 mg/dL for males and 1.4 for females, or calculated creatinine clearance less than 60 L/min.
* Males intending to impregnate others or donate sperm before, during or within 1 month after participating in the study.
* A history of cancer other than squamous or basal cell carcinoma of the skin that has not been in full remission for at least 5 years.
* A history of laser treatment for diabetic retinopathy within 6 months of screening.
* Treated for diabetic gastric paresis, gastric banding, or gastric bypass.
* New York Heart Association Class III or IV heart failure.
* History of coronary angioplasty, coronary stent placement, coronary bypass surgery, myocardial infarction, stroke or transient ischemic attack within 3 months prior to screening.
* Known history of human immunodeficiency virus, hepatitis B or C.
* Alcohol or substance abuse within 2 years prior to screening.
* Is required to take or intends to continue taking any disallowed medication, any prescription medication, herbal treatment or over-the counter medication that may interfere with evaluation of the study medication, including:

  * Any investigational drug within 30 days
  * Any investigational diabetic drug within 3 months
  * Any antidiabetic drug in the dipeptidyl peptidase-4 inhibitors or glucagon-like peptide-1 mimetics classes within 90 days prior to Screening other than metformin
  * Prior treatment with alogliptin.
  * Weight-loss drugs
  * Oral or systemically injected glucocorticoids
* A hypersensitivity allergy or anaphylactic reaction to any dipeptidyl peptidase-4 drug, metformin or glipizide.
* Has a documented history or concurrent signs of significant thyroid disease (eg, autoimmune thyroid diseases such as Graves disease and Hashimoto thyroiditis or active thyroid nodules).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2639 (Actual)
Dates: Start 2009-03; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Clinical Science, Study Director — Takeda
Locations (261):
- United States (94):
  - Montgomery, Alabama
  - Muscle Shoals, Alabama
  - Pell City, Alabama
  - Mesa, Arizona
  - Peoria, Arizona
  - Phoenix, Arizona
  - Sierra Vista, Arizona
  - Tempe, Arizona
  - Tucson, Arizona
  - Anaheim, California
  - Artesia, California
  - Chico, California
  - Los Alamitos, California
  - Mission Viejo, California
  - National City, California
  - Northridge, California
  - Pismo Beach, California
  - Riverside, California
  - Roseville, California
  - Sacramento, California
  - San Diego, California
  - Santa Monica, California
  - Tustin, California
  - Arvada, Colorado
  - Colorado Springs, Colorado
  - Ridgefield, Connecticut
  - Waterbury, Connecticut
  - Brooksville, Florida
  - New Port Richey, Florida
  - North Miami Beach, Florida
  - Ocala, Florida
  - Opa-locka, Florida
  - Orlando, Florida
  - Augusta, Georgia
  - Savannah, Georgia
  - Addison, Illinois
  - Chicago, Illinois
  - Bloomington, Indiana
  - Evansville, Indiana
  - Indianapolis, Indiana
  - Mishawaka, Indiana
  - South Bend, Indiana
  - Lexington, Kentucky
  - Munfordville, Kentucky
  - Marrero, Louisiana
  - Bangor, Maine
  - Elkridge, Maryland
  - Oxon Hill, Maryland
  - North Dartmouth, Massachusetts
  - Ann Arbor, Michigan
  - Flint, Michigan
  - Picayune, Mississippi
  - City of Saint Peters, Missouri
  - Springfield, Missouri
  - St Louis, Missouri
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Albuquerque, New Mexico
  - New Windsor, New York
  - New York, New York
  - Rochester, New York
  - Fargo, North Dakota
  - Beachwood, Ohio
  - Cincinnati, Ohio
  - Dayton, Ohio
  - Willoughby Hills, Ohio
  - Zanesville, Ohio
  - Norman, Oklahoma
  - Oklahoma City, Oklahoma
  - Medford, Oregon
  - Havertown, Pennsylvania
  - Norristown, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Tipton, Pennsylvania
  - Anderson, South Carolina
  - Charleston, South Carolina
  - Greer, South Carolina
  - Rapid City, South Dakota
  - New Tazewell, Tennessee
  - Arlington, Texas
  - Carrollton, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Hurst, Texas
  - Katy, Texas
  - San Antonio, Texas
  - Spring, Texas
  - Temple, Texas
  - Midvale, Utah
  - Hampton, Virginia
  - Lewisburg, West Virginia
  - Milwaukee, Wisconsin
- Mar del Plata, Argentina
- Australia (4):
  - Garran, Australian Capital Territory
  - Wollongong, New South Wales
  - Herston, Queensland
  - Nedlands, Western Australia
- Austria (2):
  - Graz
  - Salzburg
- Brazil (5):
  - Recife, Pernambuco
  - Brasília - DF, Planalto Central
  - Mogi das Cruzes, São Paulo
  - São Paulo, São Paulo
  - Fortaleza
- Canada (12):
  - St. John's, Newfoundland and Labrador
  - Brampton, Ontario
  - Collingwood, Ontario
  - Corunna, Ontario
  - Etobichoke, Ontario
  - Etobicoke, Ontario
  - Mississauga, Ontario
  - Smith Falls, Ontario
  - Smiths Falls, Ontario
  - Toronto, Ontario
  - Granby, Quebec
  - Montreal, Quebec
- Chile (2):
  - Providencia, Santiago Metropolitan
  - Santiago, Santiago Metropolitan
- Germany (7):
  - Potsdam, Brandenburg
  - Kelkheim, Hesse
  - Offenbach, Hesse
  - Münster, North Rhine-Westphalia
  - Mainz, Rhineland-Palatinate
  - Neuwied, Rhineland-Palatinate
  - Rhaunen, Rhineland-Palatinate
- Guatemala City, Departamento de Guatemala, Guatemala
- Hong Kong (3):
  - Kowloon, Kowloon
  - Wong Tai Sin, Kowloon
  - Pok Fu Lam, Southern District
- Hungary (9):
  - Pécs, Baranya
  - Gyula, Bekes County
  - Miskolc, Borsod-Abauj Zemplen county
  - Budapest, Budapest
  - Kalocsa, Bács-Kiskun county
  - Makó, Csongrád megye
  - Szentes, Csongrád megye
  - Nyíregyháza, Szabolcs-Szatmár-Bereg
  - Zalaegerszeg, Zala County
- India (8):
  - Hyderabad, Andhra Pradesh
  - Patna, Bihar
  - Karnāl, Haryana
  - Bangalore, Karnataka
  - Belagavi, Karnataka
  - Bhopal, Madhya Pradesh
  - Mumbai, Maharashtra
  - Trichy, Tamil Nadu
- Israel (14):
  - Kfar Saba, Center District
  - Kfar Saba, Central District
  - Matan, Central District
  - Petah Tikva, Central District
  - Hadera, Haifa District
  - Haifa, Haifa District
  - Jerusalem, Jerusalem
  - Nahariya, Northern District
  - Safed, Northern District
  - Ashkelon, Southern District
  - Beersheba, Southern District
  - Holon, Tel Aviv
  - Tel Aviv, Tel Aviv
  - Safed
- Italy (3):
  - Milan, Milan
  - Perugia, Perugia
  - Pistoia, Pistoia
- Latvia (8):
  - Daugavpils
  - Liepāja
  - Limbaži
  - Ogre
  - Riga
  - Talsi
  - Tukums
  - Valmiera
- Lithuania (7):
  - Alytus
  - Kaunas
  - Kėdainiai
  - Klaipėda
  - Palanga
  - Panevezys
  - Vilnius
- Malaysia (7):
  - Ipoh
  - Kajang
  - Kota Bharu
  - Kuala Terengganu
  - Kuantan
  - Malacca
  - Taiping
- Mexico (6):
  - Tlalnepantla, Edo de Mexico
  - Guadalajara, Jalisco
  - Mexico City, Mexico City
  - Monterrey, Nuevo León
  - Huixquilucan Edo. de Mexico
  - Mexico City
- New Zealand (8):
  - Auckland
  - Christchurch
  - Hamilton
  - Otahuhu
  - Palmerston North
  - Takapuna
  - Tauranga
  - Wellington
- Peru (3):
  - Chiclayo, Lambayeque
  - Lima, San Juan de Miraflores
  - Ica
- Manila, Philippines
- Poland (7):
  - Bytom
  - Gniewkowo
  - Krakow
  - Radom
  - Rzeszów
  - Tychy
  - Warsaw
- Puerto Rico (2):
  - Ponce
  - San Juan
- Romania (6):
  - Bacau
  - Bucharest
  - Galati
  - Oradea
  - Sibiu
  - Târgu Mureş
- Russia (7):
  - Arkhangelsk
  - Irkutsk
  - Moscow
  - Saint Petersburg
  - Samara
  - Smolensk
  - Yaroslavl
- Singapore, Singapore
- South Africa (6):
  - Port Elizabeth, Eastern Cape
  - Johannesburg, Gauteng
  - Pretoria, Gauteng
  - Durban, KwaZulu-Natal
  - Tongaat, KwaZulu-Natal
  - Cape Town, Western Cape
- South Korea (3):
  - Gwangju, Honam
  - Daejeon, Hoseo
  - Daegu, Yeongnam
- Spain (3):
  - Barcelona, Catalonia
  - Santiago de Compostela, Galicia
  - Alicante
- Thailand (4):
  - Amphure Muang
  - Bangkok
  - Chiang Mai
  - Khon Kaen
- Ukraine (10):
  - Dnepropertovsk
  - Dnipropetrovsk
  - Donetsk
  - Kharkiv
  - Kyiv
  - Lviv
  - Vinnytsa
  - Vinnytsia
  - Zaporizhye
  - Zaporizhzhya
- United Kingdom (7):
  - Aintree-Liverpool
  - Bath
  - Bournemouth
  - Dundee
  - London
  - Stevenage
  - Swansea

REFERENCES:
- [Derived] Gordon J, McEwan P, Hurst M, Puelles J. The Cost-Effectiveness of Alogliptin Versus Sulfonylurea as Add-on Therapy to Metformin in Patients with Uncontrolled Type 2 Diabetes Mellitus. Diabetes Ther. 2016 Dec;7(4):825-845. doi: 10.1007/s13300-016-0206-7. Epub 2016 Oct 27. PMID 27787778

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 310 study sites worldwide from 05 March 2009 to 17 October 2012.
Pre-assignment Details: Participants with type 2 diabetes mellitus experiencing inadequate glycemic control while on metformin therapy were enrolled equally in 1 of 3 treatment groups: alogliptin 12.5 mg once daily (QD), alogliptin 25 mg QD, and glipizide 5 mg QD.
Period: Overall Study
Arm/Group | Metformin + Alogliptin 12.5 mg | Metformin + Alogliptin 25 mg | Metformin + Glipizide
Started | 880 | 885 | 874
Received Study Drug | 873 | 878 | 869
Completed | 472 | 493 | 427
Not Completed | 408 | 392 | 447
Not completed — Hyperglycemic rescue | 231 | 201 | 235
Not completed — Adverse Event | 60 | 74 | 82
Not completed — Major protocol deviation | 24 | 16 | 15
Not completed — Lost to Follow-up | 20 | 22 | 28
Not completed — Voluntary withdrawal | 48 | 52 | 62
Not completed — Pregnancy | 1 | 2 | 0
Not completed — Investigator discretion | 9 | 8 | 10
Not completed — Other | 15 | 17 | 14
Not completed — Randomized in error | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Randomized Set included all enrolled subjects who were subsequently randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin + Alogliptin 12.5 mg | Metformin + Alogliptin 25 mg | Metformin + Glipizide | Total
Number analyzed (Participants) | 880 | 885 | 874 | 2639
Age Continuous [Mean (Standard Deviation); unit: years] | 55.2 (9.60) | 55.5 (9.81) | 55.4 (9.60) | 55.4 (9.67)
Age, Customized [Number; unit: participants] — Categories ≥65 years and ≥75 years are not mutually exclusive. Participants ≥75 years are counted in both categories.
  participants
    <65 years | 734 | 710 | 723 | 2167
    ≥65 years | 146 | 175 | 151 | 472
    ≥75 years | 13 | 17 | 15 | 45
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 461 | 433 | 433 | 1327
  Male | 419 | 452 | 441 | 1312
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 40 | 42 | 36 | 118
  Asian | 191 | 207 | 203 | 601
  Black or African American | 74 | 66 | 81 | 221
  Native Hawaiian or Other Pacific Islander | 7 | 1 | 4 | 12
  White | 557 | 555 | 533 | 1645
  Multiracial | 11 | 14 | 17 | 42
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 192 | 204 | 192 | 588
  Not Hispanic or Latino | 688 | 681 | 682 | 2051
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI data available for 879, 885 and 872 participants in each treatment arm, respectively.
  kg/m^2 | 31.27 (5.417) | 31.27 (5.341) | 31.11 (5.320) | 31.22 (5.358)
Glycosylated hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage] — Mean HbA1c data includes 877, 883 and 870 participants in each treatment arm, respectively.
  percentage | 7.59 (0.599) | 7.61 (0.606) | 7.60 (0.617) | 7.60 (0.607)
Baseline HbA1c Category [Number; unit: participants]
  <8.0% | 615 | 620 | 613 | 1848
  ≥8.0% | 265 | 265 | 261 | 791
Diabetes duration [Mean (Standard Deviation); unit: years] — Diabetes duration data available for 880, 884 and 874 participants in each treatment arm, respectively.
  years | 5.65 (5.324) | 5.42 (4.730) | 5.48 (4.884) | 5.52 (4.985)
Metformin dose [Mean (Standard Deviation); unit: mg] | 1825.2 (405.59) | 1837.2 (373.06) | 1823.4 (390.63) | 1828.6 (389.85)
Glomerular filtration rate [Mean (Standard Deviation); unit: mL/min/1.73m^2] — Glomerular filtration rate (GFR) was calculated using the modification of diet in renal disease (MDRD) formula and the Cockcroft-Gault formula. Data include 877, 883 and 870 participants in each treatment arm, respectively.
  mL/min/1.73m^2
    MDRD | 83.04 (16.586) | 82.35 (16.199) | 82.28 (16.994) | 82.56 (16.591)
    Cockcroft-Gault | 109.3 (33.40) | 109.3 (32.85) | 108.0 (32.64) | 108.9 (32.96)
Smoking history [Number; unit: participants]
  Never smoked | 543 | 586 | 578 | 1707
  Current smoker | 135 | 122 | 111 | 368
  Ex-smoker | 202 | 177 | 185 | 564

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c) at Week 52
Description: The change from Baseline to Week 52 in HbA1c (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound). The least squares (LS) means are from an analysis of covariance (ANCOVA) model with treatment, study schedule, and geographic region as class variables, and Baseline metformin dose and Baseline HbA1c as covariates.
Time Frame: Baseline and Week 52
Population: The Per-protocol set included all randomized patients who took at least 1 dose of double-blind study drug, with a Baseline assessment and at least 1 post-baseline assessment for that variable and who had no major protocol violations. Last observation carried forward (LOCF) was used.
Measure: Least Squares Mean (Standard Error); unit: percentage glycosylated hemoglobin
Arm/Group | Metformin + Alogliptin 12.5 mg | Metformin + Alogliptin 25 mg | Metformin + Glipizide
Number analyzed (Participants) | 371 | 382 | 336
percentage glycosylated hemoglobin | -0.81 (0.027) | -0.76 (0.027) | -0.73 (0.029)
Statistical Analysis 1: Comparison: Metformin + Alogliptin 25 mg vs Metformin + Glipizide; The null hypotheses were tested in a fixed order at the 1-sided 0.0125 significance level at Weeks 52 and 104, independently: H01: Alogliptin 25 mg was inferior in HbA1c change from Baseline vs glipizide. H02: Alogliptin 12.5 mg was inferior vs glipizide. H03: Alogliptin 25 mg was not superior vs glipizide. H04: Alogliptin 12.5 mg was not superior vs glipizide. Each subsequent null hypothesis was tested only if all previously tested null hypotheses were rejected with respect to Weeks 52 and 104; Test type: Non-Inferiority or Equivalence — Non-inferiority was met if the upper limit of the 1-sided 98.75% CI for the difference between alogliptin 25 mg and glipizide in HbA1c change from Baseline was less than 0.3%. If the null hypothesis H01 was rejected, then H02 was tested to show noninferiority of alogliptin 12.5 mg versus glipizide with a margin of 0.3%. Non-inferiority was met if the upper limit of the 1-sided 98.75% CI for the difference between alogliptin 12.5 mg and glipizide in HbA1c change from Baseline was less than 0.3%; LS Mean Difference = -0.03, 98.75% CI 1-sided [upper limit 0.059]
Statistical Analysis 2: Comparison: Metformin + Alogliptin 12.5 mg vs Metformin + Glipizide; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; LS Mean Difference = -0.09, 98.75% CI 1-sided [upper limit 0.003]

2. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin at Other Time Points
Description: The change from Baseline over time in HbA1c (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound). LS means are from an ANCOVA model with treatment, study schedule, and geographic region as class variables, and Baseline metformin dose and Baseline HbA1c as covariates.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, 26, 39, 65, 78, and 91.
Population: Per-protocol set; LOCF was used.
Measure: Least Squares Mean (Standard Error); unit: percentage of glycosylated hemoglobin
Arm/Group | Metformin + Alogliptin 12.5 mg | Metformin + Alogliptin 25 mg | Metformin + Glipizide
Number analyzed (Participants) | 371 | 382 | 336
percentage of glycosylated hemoglobin
  Week 4 (n=341, 354, 318) | -0.37 (0.020) | -0.40 (0.020) | -0.41 (0.021)
  Week 8 (n=370, 382, 336) | -0.56 (0.024) | -0.60 (0.024) | -0.66 (0.025)
  Week 12 (n=371, 382, 336) | -0.69 (0.025) | -0.71 (0.025) | -0.78 (0.026)
  Week 16 (n=371, 382, 336) | -0.74 (0.026) | -0.76 (0.025) | -0.78 (0.027)
  Week 20 (n=371, 382, 336) | -0.76 (0.026) | -0.78 (0.025) | -0.79 (0.027)
  Week 26 (n=371, 382, 336) | -0.80 (0.027) | -0.79 (0.026) | -0.80 (0.028)
  Week 39 (n=371, 382, 336) | -0.81 (0.026) | -0.81 (0.025) | -0.74 (0.027)
  Week 65 (n=371, 382, 336) | -0.81 (0.029) | -0.83 (0.028) | -0.76 (0.030)
  Week 78 (n=371, 382, 336) | -0.82 (0.030) | -0.80 (0.030) | -0.73 (0.032)
  Week 91 (n=371, 382, 336) | -0.76 (0.033) | -0.77 (0.033) | -0.68 (0.035)

3. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose Over Time
Description: The change from Baseline in fasting plasma glucose (FPG) was assessed at Weeks 2, 4, 8, 12, 16, 20, 26, 39, 52, 65, 78, 91, and 104. LS means are from an ANCOVA model with treatment, study schedule, and geographic region as class variables, and Baseline FPG and Baseline metformin dose as covariates.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20, 26, 39, 52, 65, 78, 91, and 104.
Population: Full analysis set, which included all randomized patients who received at least 1 dose of double-blind study drug who had a Baseline assessment and at least 1 post-baseline assessment for FPG. LOCF was used.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Metformin + Alogliptin 12.5 mg | Metformin + Alogliptin 25 mg | Metformin + Glipizide
Number analyzed (Participants) | 867 | 867 | 859
mg/dL
  Week 2 (n=781, 803, 777) | -10.2 (0.89) | -11.4 (0.87) | -7.7 (0.89)
  Week 4 (n=863, 865, 855) | -10.6 (0.85) | -11.6 (0.85) | -10.2 (0.85)
  Week 8 (n=867, 867, 859) | -9.2 (0.91) | -11.6 (0.91) | -9.3 (0.92)
  Week 12 (n=867, 867, 859) | -10.7 (0.94) | -11.2 (0.94) | -9.4 (0.95)
  Week 16 (n=867, 867, 859) | -8.6 (0.98) | -9.9 (0.98) | -7.1 (0.98)
  Week 20 (n=867, 867, 859) | -7.6 (1.02) | -10.1 (1.02) | -5.5 (1.02)
  Week 26 (n=867, 867, 859) | -7.5 (1.06) | -10.1 (1.06) | -4.3 (1.06)
  Week 39 (n=867, 867, 859) | -6.9 (1.14) | -8.4 (1.14) | -0.6 (1.15)
  Week 52 (n=867, 867, 859) | -5.0 (1.22) | -7.0 (1.22) | 0.9 (1.23)
  Week 65 (n=867, 867, 859) | -3.4 (1.21) | -5.9 (1.21) | 1.4 (1.21)
  Week 78 (n=867, 867, 859) | -2.8 (1.47) | -5.1 (1.47) | 5.1 (1.48)
  Week 91 (n=867, 867, 859) | -0.9 (1.27) | -3.4 (1.27) | 4.9 (1.28)
  Week 104 (n=867, 867, 859) | -0.9 (1.28) | -3.2 (1.28) | 5.4 (1.29)

4. Secondary Outcome: Percentage of Participants With Glycosylated Hemoglobin Less Than or Equal to 6.5%
Description: The percentage of participants with HbA1c less than or equal to 6.5% at Weeks 26, 52, 78, and 104. Participants who did not complete the scheduled Week 104 visit were assessed based on their response at the time of discontinuation.
Time Frame: Weeks 26, 52, 78, and 104.
Population: Full analysis set. Participants who did not complete the scheduled Week 26, Week 52, Week 78 or Week 104 visit were assessed based on their response at the time of discontinuation.
Measure: Number; unit: percentage of participants
Arm/Group | Metformin + Alogliptin 12.5 mg | Metformin + Alogliptin 25 mg | Metformin + Glipizide
Number analyzed (Participants) | 873 | 878 | 869
percentage of participants
  Week 26 | 25.6 | 26.2 | 24.8
  Week 52 | 24.5 | 24.8 | 20.8
  Week 78 | 24.2 | 26.4 | 21.8
  Week 104 | 23.5 | 24.1 | 19.0

5. Secondary Outcome: Percentage of Participants With Glycosylated Hemoglobin Less Than or Equal to 7.0%
Description: Percentage of participants with HbA1c ≤ 7.0% at Weeks 26, 52, 78, and 104. Participants who did not complete the scheduled Week 104 visit were assessed based on their response at the time of discontinuation.
Time Frame: Weeks 26, 52, 78, and 104.
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Metformin + Alogliptin 12.5 mg | Metformin + Alogliptin 25 mg | Metformin + Glipizide
Number analyzed (Participants) | 873 | 878 | 869
percentage of participants
  Week 26 | 56.4 | 59.2 | 56.1
  Week 52 | 51.7 | 55.5 | 47.4
  Week 78 | 48.8 | 52.4 | 46.6
  Week 104 | 45.6 | 48.5 | 42.8

6. Secondary Outcome: Change From Baseline in Body Weight Over Time
Description: LS Means are from an ANCOVA model with treatment, study schedule and geographic region as class variables, and Baseline weight and Baseline metformin dose as covariates.
Time Frame: Baseline and Weeks 12, 26, 39, 52, 65, 78, 91, and 104.
Population: Full analysis set, LOCF was used.
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Metformin + Alogliptin 12.5 mg | Metformin + Alogliptin 25 mg | Metformin + Glipizide
Number analyzed (Participants) | 867 | 868 | 861
kg
  Week 12 | -0.51 (0.076) | -0.53 (0.076) | 0.71 (0.077)
  Week 26 | -0.65 (0.101) | -0.71 (0.101) | 0.86 (0.101)
  Week 39 | -0.60 (0.109) | -0.86 (0.109) | 0.97 (0.110)
  Week 52 | -0.63 (0.117) | -0.90 (0.117) | 0.89 (0.117)
  Week 65 | -0.70 (0.122) | -0.92 (0.122) | 0.87 (0.123)
  Week 78 | -0.78 (0.124) | -0.94 (0.124) | 0.88 (0.125)
  Week 91 | -0.67 (0.127) | -0.88 (0.127) | 0.89 (0.127)
  Week 104 | -0.68 (0.127) | -0.89 (0.127) | 0.95 (0.127)

7. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c) at Week 104
Description: The change from Baseline to Week 104 in HbA1c (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound). The least squares (LS) means are from an analysis of covariance (ANCOVA) model with treatment, study schedule, and geographic region as class variables, and Baseline metformin dose and Baseline HbA1c as covariates.
Time Frame: Baseline and Week 104
Population: The Per-protocol set included all randomized patients who took at least 1 dose of double-blind study drug, with a Baseline assessment and at least 1 post-baseline assessment for that variable and who had no major protocol violations. Last observation carried forward was used (LOCF).
Measure: Least Squares Mean (Standard Error); unit: percentage glycosylated hemoglobin
Arm/Group | Metformin + Alogliptin 12.5 mg | Metformin + Alogliptin 25 mg | Metformin + Glipizide
Number analyzed (Participants) | 371 | 382 | 336
percentage glycosylated hemoglobin | -0.68 (0.037) | -0.72 (0.037) | -0.59 (0.039)
Statistical Analysis 1: Comparison: Metformin + Alogliptin 25 mg vs Metformin + Glipizide; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; LS Mean Difference = -0.13, 98.75% CI 1-sided [upper limit -0.006]
Statistical Analysis 2: Comparison: Metformin + Alogliptin 12.5 mg vs Metformin + Glipizide; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; LS Mean Difference = -0.09, 98.75% CI 1-sided [upper limit 0.035]

ADVERSE EVENTS:
Time Frame: Collection of adverse events commenced from the time the participant was first administered double-blind study medication until the end of the study and from spontaneous reporting for 30 days after the end of treatment (up to 108 weeks).
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Metformin + Alogliptin 12.5 mg | Metformin + Alogliptin 25 mg | Metformin + Glipizide
Serious Adverse Events (participants affected / at risk) | 86/873 | 97/878 | 81/869
Other Adverse Events (participants affected / at risk) | 688/873 | 687/878 | 668/869
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Metformin + Alogliptin 12.5 mg (N=873) | Metformin + Alogliptin 25 mg (N=878) | Metformin + Glipizide (N=869)
Coronary artery disease (Cardiac disorders) | 5 | 3 | 2
Angina unstable (Cardiac disorders) | 1 | 4 | 4
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 5
Atrial fibrillation (Cardiac disorders) | 1 | 3 | 2
Atrial flutter (Cardiac disorders) | 2 | 2 | 1
Cardiac failure (Cardiac disorders) | 0 | 3 | 1
Cardiac failure congestive (Cardiac disorders) | 2 | 1 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1 | 3
Angina pectoris (Cardiac disorders) | 0 | 2 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 2
Atrioventricular block complete (Cardiac disorders) | 1 | 0 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 1 | 1
Silent myocardial infarction (Cardiac disorders) | 0 | 2 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1 | 0
Atrioventricular block (Cardiac disorders) | 0 | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 0
Congestive cardiomyopathy (Cardiac disorders) | 0 | 1 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 1 | 0
Left ventricular failure (Cardiac disorders) | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0
Right ventricular failure (Cardiac disorders) | 1 | 0 | 0
Tachyarrhythmia (Cardiac disorders) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 3 | 1 | 3
Pneumonia (Infections and infestations) | 1 | 2 | 2
Gastroenteritis (Infections and infestations) | 2 | 2 | 0
Dengue fever (Infections and infestations) | 1 | 0 | 2
Diverticulitis (Infections and infestations) | 1 | 1 | 1
Hepatitis viral (Infections and infestations) | 1 | 0 | 2
Urinary tract infection (Infections and infestations) | 1 | 1 | 1
Urosepsis (Infections and infestations) | 0 | 1 | 1
Abdominal abscess (Infections and infestations) | 0 | 0 | 1
Abscess limb (Infections and infestations) | 0 | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 1
Amoebiasis (Infections and infestations) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1
Cystitis (Infections and infestations) | 1 | 0 | 0
Gangrene (Infections and infestations) | 0 | 1 | 0
Gastroenteritis salmonella (Infections and infestations) | 0 | 1 | 0
Lobar pneumonia (Infections and infestations) | 0 | 1 | 0
Malaria (Infections and infestations) | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 1 | 0 | 0
Pneumocystis jiroveci pneumonia (Infections and infestations) | 0 | 0 | 1
Scrotal abscess (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 1 | 3
Syncope (Nervous system disorders) | 2 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 0 | 1
Headache (Nervous system disorders) | 1 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 2 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0
Haemorrhagic stroke (Nervous system disorders) | 1 | 0 | 0
Intercostal neuralgia (Nervous system disorders) | 0 | 1 | 0
Neuralgia (Nervous system disorders) | 1 | 0 | 0
Parkinsonism (Nervous system disorders) | 0 | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0
Radiculopathy (Nervous system disorders) | 0 | 1 | 0
Tension headache (Nervous system disorders) | 1 | 0 | 0
VIIth nerve paralysis (Nervous system disorders) | 1 | 0 | 0
VIth nerve paralysis (Nervous system disorders) | 0 | 0 | 1
Vertebrobasilar insufficiency (Nervous system disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 3 | 4
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myalgia intercostal (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Polymyositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 2 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 2
Inguinal hernia (Gastrointestinal disorders) | 1 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 1 | 1
Anal fistula (Gastrointestinal disorders) | 1 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 0 | 1
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1
Umbilical hernia, obstructive (Gastrointestinal disorders) | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Colon cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Non-small cell lung cancer stage IIIB (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Renal oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 2 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 2
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 1
Comminuted fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Peripheral nerve injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 2 | 3
Nephrolithiasis (Renal and urinary disorders) | 2 | 2 | 0
Renal colic (Renal and urinary disorders) | 1 | 1 | 1
Calculus urinary (Renal and urinary disorders) | 0 | 1 | 0
Diabetic nephropathy (Renal and urinary disorders) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 3 | 0
Hypertensive crisis (Vascular disorders) | 0 | 2 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 1 | 0
Aortic aneurysm (Vascular disorders) | 1 | 0 | 0
Arterial thrombosis limb (Vascular disorders) | 1 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 1
Femoral artery occlusion (Vascular disorders) | 0 | 0 | 1
Iliac artery occlusion (Vascular disorders) | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 3 | 4 | 3
Chest pain (General disorders) | 0 | 2 | 0
Hernia (General disorders) | 0 | 1 | 0
Sudden death (General disorders) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Granulomatous pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 1 | 0
Adenomyosis (Reproductive system and breast disorders) | 1 | 0 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 0 | 0
Cervix disorder (Reproductive system and breast disorders) | 1 | 0 | 0
Cystocele (Reproductive system and breast disorders) | 1 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 0
Epididymitis (Reproductive system and breast disorders) | 1 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0
Rectocele (Reproductive system and breast disorders) | 1 | 0 | 0
Uterine prolapse (Reproductive system and breast disorders) | 1 | 0 | 0
Uterovaginal prolapse (Reproductive system and breast disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 1 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 3 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0 | 0
Cataract (Eye disorders) | 1 | 1 | 1
Cataract nuclear (Eye disorders) | 1 | 0 | 0
Cataract subcapsular (Eye disorders) | 1 | 0 | 0
Iridocyclitis (Eye disorders) | 0 | 0 | 1
Retinal detachment (Eye disorders) | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0
Bipolar disorder (Psychiatric disorders) | 1 | 0 | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 1 | 0
Depressed mood (Psychiatric disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
Schizophrenia (Psychiatric disorders) | 0 | 0 | 1
Acute vestibular syndrome (Ear and labyrinth disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Vertigo positional (Ear and labyrinth disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Primary hyperaldosteronism (Endocrine disorders) | 0 | 0 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0
Abortion (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Metformin + Alogliptin 12.5 mg (N=873) | Metformin + Alogliptin 25 mg (N=878) | Metformin + Glipizide (N=869)
Diarrhoea (Gastrointestinal disorders) | 60 | 60 | 63
Upper respiratory tract infection (Infections and infestations) | 84 | 90 | 76
Nasopharyngitis (Infections and infestations) | 78 | 67 | 61
Anaemia (Blood and lymphatic system disorders) | 16 | 37 | 32
Nausea (Gastrointestinal disorders) | 28 | 32 | 20
Fatigue (General disorders) | 20 | 19 | 28
Asthenia (General disorders) | 14 | 15 | 27
Influenza (Infections and infestations) | 36 | 36 | 42
Urinary tract infection (Infections and infestations) | 41 | 33 | 38
Bronchitis (Infections and infestations) | 39 | 36 | 36
Sinusitis (Infections and infestations) | 26 | 29 | 23
Creatinine renal clearance decreased (Investigations) | 23 | 34 | 32
Hypoglycaemia (Metabolism and nutrition disorders) | 18 | 6 | 91
Dyslipidaemia (Metabolism and nutrition disorders) | 22 | 20 | 34
Back pain (Musculoskeletal and connective tissue disorders) | 54 | 45 | 49
Arthralgia (Musculoskeletal and connective tissue disorders) | 38 | 42 | 40
Pain in extremity (Musculoskeletal and connective tissue disorders) | 28 | 28 | 33
Headache (Nervous system disorders) | 45 | 60 | 46
Dizziness (Nervous system disorders) | 24 | 24 | 29
Tremor (Nervous system disorders) | 5 | 3 | 29
Cough (Respiratory, thoracic and mediastinal disorders) | 35 | 26 | 33
Hypertension (Vascular disorders) | 45 | 67 | 65

LIMITATIONS AND CAVEATS:
The Week 52 results summarized in herein differ from the Week 52 results summarized in an interim analysis, because the per protocol set (PPS) defined for the final analysis included fewer subjects than the PPS defined for the interim analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.